CLINICAL TRIAL: NCT06261593
Title: Efficacy of a Physiotherapy Intervention Through Blood Flow Restriction in Improving Muscle Strength in Patients With Hemophilic Ankle Arthropathy: Multicenter Randomized Clinical Study
Brief Title: Blood Flow Restriction in Improving Muscle Strength of Patients With Hemophilic Ankle Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ankle-Blood
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia
Keywords: Hemophilia; Blood flow restriction; Physiotherapy; Muscular strength; Muscle activation; Range of Motion; Chronic pain; Stability
MeSH Terms: conditions — Hemophilia A; Chronic Pain | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention will consist of carrying out a physiotherapy protocol, consisting of strength training through blood flow restriction, with an occlusion pressure of 40-50% of the LOP (Limb Occlusion Pressure) and a load of 20-30%. of 1RM performed ad hoc for patients with hemophilic arthropathy.
  The intervention protocol will be carried out in person under the supervision of the main researcher. The intervention will last 4 weeks, with a frequency of 3 weekly sessions. In total there will be 12 sessions lasting approximately 30-45 minutes.
  Interventions: Other: Blood flow restriction
- Control group (No Intervention): The patients included in the control group will not receive any Physiotherapy intervention and will continue with their usual routine, being evaluated in the same periods as the rest of the patients

INTERVENTIONS:
Other: Blood flow restriction — The intervention protocol through blood flow restriction in patients with hemophilic arthropathy will consist of performing two exercises: heel elevation and ankle dorsiflexion in a closed kinetic chain. Both exercises will be performed for 5-10 minutes, performing 4 series (30, 15, 15, 15 repetitions) with 30 seconds of rest between series
  Arms: Experimental group

SUMMARY:
Background. The main physical sequela of patients with hemophilia is the development of a progressive, degenerative intra-articular lesion, known as hemophilic arthropathy). This sequela is manifested by chronic pain, limited range of motion, axial abnormalities, and periarticular muscle atrophy.

Objective. To assess the safety and effectiveness of an intervention through blood flow restriction, regarding the frequency of bleeding and the improvement in muscle activation and strength, range of motion, stability, joint pain, joint status and the perception of quality of life in patients with hemophilic ankle arthropathy.

Study design. Randomized, multicenter, single-blind clinical study. Method. 32 patients with hemophilia A and B will be recruited in this study. Patients will be recruited in 4 regions of Spain. The dependent variables will be: bleeding frequency (self-registration), pain (measured with the visual analog scale and pressure algometer), quality of life (SF-36 scale), joint status (Hemophilia Joint Health Score scale), strength (dynamometer) and muscle activation (surface electromyograph), range of motion (goniometer) and stability (The Single Leg Stance Test). Three evaluations will be carried out: pre-treatment, post-treatment and after a follow-up period of 4 weeks.

Expected results. Observe the safety of blood flow restriction in hemophilia patients. To analyze the efficacy of blood flow restriction in improving muscle strength and activation, range of motion, chronic pain, stabilit, and the perception of quality of life in patients with hemophilic ankle arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* People with a medical diagnosis of hemophilic ankle arthropathy
* Patients over 18 years of age
* Paceinets in prophylactic or on-demand treatment regimen with FVIII/FIX concentrates.
* Failure to sign the informed consent document

Exclusion Criteria:

* Patients with neurological or cognitive alterations that prevent understanding of the questionnaires
* Amputee patients, epileptics or patients with severe vision problems
* Patients who are receiving physiotherapy treatment at the time of the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-04-06 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline hemarthrosis after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  A self-registration will be used to evaluate the frequency of bleeding, and thus the safety of the technique. This selfregistration will be given to each patient at the beginning of the study and they must fill in the number of hemarthrosis and their main characteristics: date, origin (traumatic or spontaneous) and location (knee, ankle or elbow). The selfregistration will be delivered to the evaluator in each of the study evaluations (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline pressure pain threshold after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With a pressure algometer (model Wagner FPN100) the investigators will measure the pressure pain threshold, at the joint level and at a distance (in another part of the body). This device measures in Newton / cm2 the pressure at which the subject perceives pain under pressure. A pressure will be made on the chosen point, which the investigators will increase at an approximate speed of 50kPa / s until the patient warns us that the sensation begins to be painful.
Change from baseline muscle strength after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With a pressure dynamometer (microFET®2 Digital Handheld model) the investigators will measure the strength of the tibialis and gastrocnemius. This device measures in Newton the force that the patient exerts in the requested muscular action. The higher the value, the greater the muscle strength. The investigators will carry out the measurements bilaterally. The patient will be asked 4 maximum isometric contractions of 5 seconds, with a rest of 30 seconds between them, against the dynamometer located in the hand of the evaluator
Change from baseline electrical activity of the muscles after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Using surface electromyography (model SHIMMMER2, Shimmer, Ireland), the investigators will evaluate the electrical activity of the musculature and its level of activation. The placement of the electrodes will be marked on the standing subjects, and they will be placed following the European recommendations for the use of the SEMG. A bipolar SEMG system will be used with circular electrodes 10 mm in diameter, 20 mm apart, placed longitudinally, in the direction of the fibers of the studied muscle, and with a remote reference electrode.
Change from baseline joint status after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With the Hemophilia Joint Health Score scale, specific for its use in patients with hemophilia, the joint status of patients with hemophilic arthropathy will be evaluated. It evaluates 8 items: inflammation and duration of this, pain, muscle atrophy and strength, crackles, and loss of flexion and extension. It has a score of 0 (no joint damage) to 20 points (maximum joint damage) per joint (elbows, knees and ankles). A gait rating is added to the 120 points (range 0-4 points), the maximum rating on this scale being 124 points
Change from baseline balance after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  With the Single Leg Stance Test, static postural control and balance will be evaluated. To perform this test, the subject must place both hands on the hips and flex the knee of the non-tested leg, leaving the opposite foot as the only support. The time will be timed (in seconds) from the moment the participant flexes his leg until he places it on the ground again or his hands come off his hips, with a maximum of 60 seconds. This test will be performed with visual support (eyes open) and without it (eyes closed). The longer the time, the better stability. The participants in this study will perform the test twice with each leg, with the best score recorded in the data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No